CLINICAL TRIAL: NCT06878989
Title: Adaptation of Human Brown Adipose Tissue to Calorie Restriction (BATON)
Brief Title: Adaptation of Human Brown Adipose Tissue to Calorie Restriction
Acronym: BATON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Hospital Clinico Universitario San Cecilio (Other); University Hospital Virgen de las Nieves (Other)
Responsible Party: Principal Investigator, Guillermo Sanchez Delgado, Ramon y Cajal Researcher, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GSD-2024-004; PID2021-127582OA-I00 (Other: University of Granada)
Record Dates: First submitted 2025-02-12; First posted 2025-03-17 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Obesity and Overweight
Keywords: Energy metabolism; Metabolic Health; Brown adipose tissue (BAT); Thermogenesis; Obesity
MeSH Terms: conditions — Obesity; Overweight | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight loss group (Experimental)
  Interventions: Behavioral: Caloric restriction diet
- Control group (Experimental)
  Interventions: Behavioral: Weight maintenance diet

INTERVENTIONS:
Behavioral: Caloric restriction diet — Dietary intervention consisting on a meal plan designed to induce an 8-10% weight loss over a 12-16 week period.
  Arms: Weight loss group
Behavioral: Weight maintenance diet — Dietary intervention consisting on a meal plan designed to maintain a stable body weight for up to 16 weeks.
  Arms: Control group

SUMMARY:
The BATON study investigates how human brown adipose tissue (BAT) adapts to a controlled caloric restriction diet in young adults with obesity. A weight maintenance diet group will be compared to a group following a diet designed to induce an 8-10% weight loss over a 12-16 week period. Outcome assessments will include advanced technologies such as PET-CT and molecular analyses of BAT. The overarching goal is to gain a deeper understanding of the role of human BAT on the regulation of body weight.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 27-40 kg/m², with a body fat percentage (determined by DXA, Hologic Wi) exceeding 25% in men and 30% in women.
* Reported stable body weight over the preceding 3 months (body weight changes of less than 3%).
* Laboratory safety test results (general biochemistry and complete blood count) within the normal reference range or with abnormalities deemed clinically insignificant by the medical research team and not requiring pharmacological treatment.
* Adequate venous access for blood sampling required by the procedures described in this protocol and absence of needle, blood, or medical procedure phobia.
* Readiness and ability to consume all foods included in the assessments and dietary intervention.
* Ability to understand and comply with study procedures, as assessed by the research team.
* Availability to participate in the study.
* Commitment to completing the study regardless of the assigned group.

Exclusion Criteria:

* Diagnosis or presence of signs or symptoms that, in the opinion of the research team, may contraindicate the dietary intervention or any of the procedures included in the study.
* Diagnosis or history of metabolic (including any type of diabetes mellitus), hematologic, pulmonary, cardiovascular, gastrointestinal, neurological, immune, hepatic, renal, urologic, or psychiatric diseases that could interfere with study outcomes or protocol adherence.
* History of any surgical procedure that, in the opinion of the research team, could alter energy metabolism or digestive function during the course of the study.
* Having been exposed to medical procedures involving an estimated radiation dose exceeding 5 mSv in the past 5 years or 10 mSv over a lifetime.
* Use of medications or supplements that are known to alter body weight or appetite.
* Weight loss exceeding 10% in the past two years or more than 5% in the past six months, unless completed weight recovery has occurred.
* Adherence to unconventional dietary patterns, such as vegan or fasting diets, or inability to tolerate the foods provided during the study.
* Pregnancy, plans to become pregnant within the next two years, postpartum period (within 12 months after delivery), or lactation.
* Perimenopausal status, defined as the presence of irregular menstrual cycles, hormonal changes indicative of perimenopause, or menopausal symptoms.
* Participation in any type of nutritional intervention or treatment within the past three months.
* Diagnosis or risk factors for the development of an eating disorder.
* Frequent disruptions in the sleep-wake cycle.
* Clinically significant abnormalities in gastric emptying, current diagnosis of any form of diabetes, blood pressure exceeding 160/90 mmHg, or resting heart rate below 50 or above 100 beats per minute (while seated), regardless of stable antihypertensive medication use.
* Active or untreated malignant disease or remission from a clinically significant malignant disease for less than five years prior to the evaluation.
* History of drug or alcohol abuse or a positive drug test, unless due to a medication prescribed by a healthcare professional.
* Smoking, vaping, or habitual use of tobacco products, unless abstinent for at least 72 consecutive hours during the past four weeks.
* Habitual caffeine consumption exceeding the equivalent of three espresso coffees per day (225 mg/day).
* Being a direct relative or household member of the research team personnel.
* Any other condition that, in the opinion of the research team, contraindicates study participation.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
BAT volume | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
BAT 18F-FDG uptake upon cold exposure | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
BAT UCP-1 protein content | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Mean adipocyte size | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).

SECONDARY OUTCOMES:
BAT transcriptomics (RNA sequencing) | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Weight (kg) | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
Waist circumference (cm) | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
Hip circumference (cm) | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
Resting Systolic blood pressure (mmHg) | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
Resting Diastolic blood pressure (mmHg) | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
Fat mass (kg) by DXA | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
Fat free mass (kg) by DXA | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
Fat mass (kg) by Bioimpedanciometry | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
Fat free mass (kg) by Bioimpedanciometry | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
Body Mass Index (kg/m2) | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
Resting Energy Expenditure (kcal/day) measured by indirect calorimetry | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
Ad libitum energy intake (kcal) measured in a test meal | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Meal-induced thermogenesis (% of resting energy expenditure) measured by indirect calorimetry | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Resting heart rate variability | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
  RMSSD, SDNN
Maximal fat oxidation (g/min) by indirect calorimetry | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Physical activity (counts) measured by accelerometry | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Sedentary time (min) measured by accelerometry | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Habitual food consumption collected by a food frequency questionnaire | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
Serum total cholesterol (mg/dl) | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Serum C-reactive protein (mg/l) | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Serum thyrotropin (µU/mL) | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Serum alanine aminotransferase (U/L) | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Serum aspartate aminotransferase (U/L) | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Serum gamma-glutamyl transferase (U/L) | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Serum triglycerides (mg/dl) | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Serum LDL cholesterol (mg/dL) | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Serum HDL cholesterol (mg/dl) | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Serum glucose (mg/dl) | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Serum insulin (U/ml) | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Serum hemoglobin A1c (mmol/mol) | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Serum triiodothyronine (ng/dL) | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Serum thyroxine (ng/dL) | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Sleep time (min) measured by accelerometry | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Handgrip strength (kg) measured using a dynamometer | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Meal-induced changes in insulin concentration (U/ml) in response to a standardized meal | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Meal-induced changes in glucose concentration (mmol/L) in response to a standardized meal | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Meal-induced changes in lactate concentrations (mmol/l) in response to a standardized meal | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Meal-induced changes in triglycerides concentrations (mg/dl) in response to a standardized meal | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Meal-induced changes in total cholesterol concentrations (mg/dL) in response to a standardized meal | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Meal-induced changes in free fatty acids (mmol/L) in response to a standardized meal | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Meal-induced changes in glycerol concentrations (mmol/l) in response to a standardized meal | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Meal-induced changes in 3-hydroxybutyrate concentrations (mmol/L) in response to a standardized meal | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Functional mobility measured by "Timed Up and Go (TUG)" test | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Walking speed (m/s) measured by a gait speed test | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Independence in activities of daily living (ADL) measured by "Barthel Index" | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Food cravings measured using the "Food Craving Inventory" questionnaire | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
Control of eating behavior measured using the "Control of Eating Weekly Questionnaire" | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
Cognitive restriction of food intake measured using the "Three-Factor Eating Questionnaire" | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
Food disinhibition measured using the "Three-Factor Eating Questionnaire" | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
Subjective hunger measured using the "Three-Factor Eating Questionnaire" | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
Binge eating behavior measured using the "Binge Eating Questionnaire" | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
Fasting appetite-related sensations measured using "Visual Analogue Scales (VAS)" | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
  The scales range from 0 to 100
Meal-induced changes in appetite-related sensations measured using "Visual Analogue Scales (VAS)" in response to a standardized meal | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
  The scales range from 0 to 100
Energy efficiency (W/Kcal) while cycling, assessed by indirect calorimetry | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Vastus lateralis thickness (cm) measured by ultrasound | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Subcutaneous fat thickness (cm) measured by ultrasound | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Superficial fat thickness (cm) measured by ultrasound | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Preperitoneal fat thickness (cm) measured by ultrasound | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss).
Carbohydrate intake (g/day) collected through three 24-hour recalls | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
Fat intake (g/day) collected through three 24-hour recalls | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
Protein intake (g/day) collected through three 24-hour recalls | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention
Fiber intake (g/day) collected through three 24-hour recalls | Baseline; End of the dietary intervention (Week 12/16, depending on when the participant achieves an 8-10% weight loss); 6 months after the end of dietary intervention; 12 months after the end of dietary intervention

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Sanchez Delgado, Ramon y Cajal Researcher, Principal Investigator — Universidad de Granada
Locations (1):
- Department of Physiology, Faculty of Medicine, University of Granada., Granada, Granada, Spain